CLINICAL TRIAL: NCT04610580
Title: A Phase 1, Randomized, 2-period, 2-sequence, Crossover With Parallel-group Extension, Open-label Study to Compare the Relative Bioavailability of 2 Oral Formulations of ALXN1840 in Healthy Adult Participants
Brief Title: Bioavailability Study of 2 Oral Formulations of ALXN1840
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1840-HV-109
Record Dates: First submitted 2020-10-13; First posted 2020-10-30 (Actual); Results first posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2023-04

CONDITIONS: Healthy
Keywords: Bioavailability; Healthy

STUDY DESIGN:
Intervention Model Description: This is a 2-period, 2-sequence, crossover study with a parallel group extension.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Crossover ALXN1840 Sequence 1 (Experimental): Participants will first receive a single dose of ALXN1840 test formulation on Day 1 of Period 1. After a washout period of 14 days, they will then receive a single dose of ALXN1840 reference formulation on Day 1 of Period 2.
  Interventions: Drug: ALXN1840
- Crossover ALXN1840 Sequence 2 (Experimental): Participants will first receive a single dose of ALXN1840 reference formulation on Day 1 of Period 1. After a washout period of 14 days, they will then receive a single dose of ALXN1840 test formulation on Day 1 of Period 2.
  Interventions: Drug: ALXN1840
- Parallel Dose-proportionality Extension: ALXN1840 Dose 1 (Experimental): Participants will receive a single dose of ALXN1840.
  Interventions: Drug: ALXN1840
- Parallel Dose-proportionality Extension: ALXN1840 Dose 2 (Experimental): Participants will receive a single dose of ALXN1840.
  Interventions: Drug: ALXN1840
- Parallel Dose-proportionality Extension: ALXN1840 Dose 3 (Experimental): Participants will receive a single dose of ALXN1840.
  Interventions: Drug: ALXN1840
- Parallel Dose-proportionality Extension: ALXN1840 Dose 4 (Experimental): Participants will receive a single dose of ALXN1840.
  Interventions: Drug: ALXN1840

INTERVENTIONS:
Drug: ALXN1840 — ALXN1840 will be administered orally.
  Other Names: Tiomolibdate choline; Tiomolibdic acid

SUMMARY:
The study will assess the relative bioavailability of 2 different formulations of ALXN1840 in healthy participants.

DETAILED DESCRIPTION:
This is a two-way crossover study consisting of 2 dosing periods assessing a test and reference formulation of ALXN1840. A dose-proportionality parallel group design extension period will be conducted following completion of the two-way crossover period of the study and will assess 5 different ascending doses of ALXN1840. There will be at least a 14-day washout following doses between Periods 1 and 2 and also at least a 14-day washout following the dose in Period 2 and the following dose in the Dose-Proportionality Extension Period.

Safety will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant history or presence of electrocardiogram findings
* Body weight ≥50 to ≤100 kilograms (kg) and body mass index 18 to <32 kg/meter squared for all participants
* Willing and able to follow protocol-specified contraception requirements

Exclusion Criteria:

* History or presence of clinical and/or laboratory disorders
* Abnormal blood pressure, defined as supine blood pressure ≤90/60 millimeters of mercury (mmHg) or >140/90 mmHg
* Lymphoma, leukemia, or any malignancy within the past 5 years
* Alanine aminotransferase, aspartate aminotransferase, or total bilirubin > upper limit of normal
* Serum copper or serum ceruloplasmin below lower limit of normal
* Hemoglobin <130 grams (g)/liter (L) for males and hemoglobin <115 g/L for females
* Significant allergies
* Smoker

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-01-31 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene S. Swenson, MD, PhD, Study Director — Alexion Pharmaceuticals, Inc.; Masood Sadaat, MD, MSc, Study Chair — Alexion Pharmaceuticals, Inc.
Locations (1):
- Nucleus Network Pty Ltd., Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included a 2-way crossover period and a dose-proportionality extension period. Participants were randomized to 1 of the 2 treatment sequences (A-B) or (B-A) in crossover period with washout between. Participants were scheduled to receive either treatment A or B on Day 1 of each dosing period. After a 14-day washout period, participants were rerandomized in dose-proportionality extension period to receive treatment C, D, E, or F.
Groups:
- Crossover: ALXN1840 Test Formulation (Treatment A) First, Then Reference Formulation (Treatment B): Participants received a single dose of ALXN1840 test formulation (15 milligrams [mg]; 12 × 1.25 mg enteric-coated [EC] mini-tablets) orally on Day 1 of the first dosing period. Then, participants received a single dose of ALXN1840 reference formulation (15 mg EC tablet) orally on Day 1 of the second dosing period.
  There was a 14-day washout between the two dosing periods.
- Crossover: ALXN1840 Reference Formulation (Treatment B) First, Then Test Formulation (Treatment A): Participants received a single dose of ALXN1840 reference formulation (15 mg EC tablet) orally on Day 1 of the first dosing period. Then, participants received a single dose of ALXN1840 test formulation (15 mg; 12 × 1.25 mg EC mini-tablets) orally on Day 1 of second dosing period.
  There was a 14-day washout between the two dosing periods.
- Dose-proportionality Extension: ALXN1840 2.5 mg (Treatment C): Participants received a single dose of ALXN1840 2.5 mg (2 × 1.25 mg EC mini-tablets) orally on Day 1.
- Dose-proportionality Extension: ALXN1840 5 mg (Treatment D): Participants received a single dose of ALXN1840 5 mg (4 × 1.25 mg EC mini-tablets) orally on Day 1.
- Dose-proportionality Extension: ALXN1840 10 mg (Treatment E): Participants received a single dose of ALXN1840 10 mg (8 × 1.25 mg EC mini-tablets) orally on Day 1.
- Dose-proportionality Extension: ALXN1840 30 mg (Treatment F): Participants received a single dose of ALXN1840 30 mg (24 × 1.25 mg EC mini-tablets) orally on Day 1.
Period: Two-way Crossover Period
Arm/Group | Crossover: ALXN1840 Test Formulation (Treatment A) First, Then Reference Formulation (Treatment B) | Crossover: ALXN1840 Reference Formulation (Treatment B) First, Then Test Formulation (Treatment A) | Dose-proportionality Extension: ALXN1840 2.5 mg (Treatment C) | Dose-proportionality Extension: ALXN1840 5 mg (Treatment D) | Dose-proportionality Extension: ALXN1840 10 mg (Treatment E) | Dose-proportionality Extension: ALXN1840 30 mg (Treatment F)
Started | 24 | 24 | 0 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug | 24 | 24 | 0 | 0 | 0 | 0
Completed | 22 | 22 | 0 | 0 | 0 | 0
Not Completed | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other than specified | 0 | 1 | 0 | 0 | 0 | 0
Period: Washout Before Extension Period
Arm/Group | Crossover: ALXN1840 Test Formulation (Treatment A) First, Then Reference Formulation (Treatment B) | Crossover: ALXN1840 Reference Formulation (Treatment B) First, Then Test Formulation (Treatment A) | Dose-proportionality Extension: ALXN1840 2.5 mg (Treatment C) | Dose-proportionality Extension: ALXN1840 5 mg (Treatment D) | Dose-proportionality Extension: ALXN1840 10 mg (Treatment E) | Dose-proportionality Extension: ALXN1840 30 mg (Treatment F)
Started | 22 | 22 | 0 | 0 | 0 | 0
Completed | 22 | 19 | 0 | 0 | 0 | 0
Not Completed | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Other than specified | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0 | 0 | 0
Period: Dose-Proportionality Extension Period
Arm/Group | Crossover: ALXN1840 Test Formulation (Treatment A) First, Then Reference Formulation (Treatment B) | Crossover: ALXN1840 Reference Formulation (Treatment B) First, Then Test Formulation (Treatment A) | Dose-proportionality Extension: ALXN1840 2.5 mg (Treatment C) | Dose-proportionality Extension: ALXN1840 5 mg (Treatment D) | Dose-proportionality Extension: ALXN1840 10 mg (Treatment E) | Dose-proportionality Extension: ALXN1840 30 mg (Treatment F)
Started | 0 | 0 | 10 | 11 | 9 | 11
Received at Least 1 Dose of Study Drug | 0 | 0 | 10 | 11 | 9 | 11
Completed | 0 | 0 | 10 | 11 | 8 | 11
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Set included all participants who received at least 1 dose of ALXN1840.
Groups:
- Overall Population: Crossover: Participants first received a single dose of ALXN1840 test formulation (15 mg; 12 × 1.25 mg EC mini-tablets) orally on Day 1 of Period 1 and then after a washout period of 14 days, received a single dose of ALXN1840 reference formulation (15 mg EC tablet) orally on Day 1 of Period 2. Dose-proportionality extension: Participants received a single dose of ALXN1840 2.5, 5, 10, or 30 mg orally on Day 1.
Arm/Group | Overall Population
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (7.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 19
  Race: Black or African American | 3
  Race: White | 24
  Race: Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Two-way Crossover Period: Maximum Observed Concentration (Cmax) For Plasma Total Molybdenum (Mo)
Description: Whole blood samples were collected for the measurement of plasma concentrations of total Mo via inductively coupled plasma-mass spectroscopy (ICP-MS).
Time Frame: predose (0.5 hour) and up to 336 hours postdose
Population: The Pharmacokinetic/Pharmacodynamic Set for the Two-way Crossover Periods (PKDS-CO) included all participants who received at least 1 dose of ALXN1840 in the Two-way Crossover Periods and had evaluable pharmacokinetic (PK) data for total and/or plasma ultrafiltrate (PUF) Mo (as surrogate measures of ALXN1840 PK) in plasma. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms (ng)/milliliter (mL)
Groups:
- Crossover: ALXN1840 Test Formulation (Treatment A): Participants received a single dose of ALXN1840 test formulation (15 mg; 12 × 1.25 mg EC mini-tablets) orally on Day 1 of each dosing period in a crossover design.
- Crossover: ALXN1840 Reference Formulation (Treatment B): Participants received a single dose of ALXN1840 reference formulation (15 mg EC tablet) orally on Day 1 of each dosing period in a crossover deign.
Arm/Group | Crossover: ALXN1840 Test Formulation (Treatment A) | Crossover: ALXN1840 Reference Formulation (Treatment B)
Number analyzed (Participants) | 45 | 46
nanograms (ng)/milliliter (mL) | 227.0186 (47.5) | 238.2725 (30.8)
Statistical Analysis 1: Comparison: Crossover: ALXN1840 Test Formulation (Treatment A) vs Crossover: ALXN1840 Reference Formulation (Treatment B); The formulation impact (12 × 1.25 mg EC mini-tablet versus 1 × 15 mg EC tablet) on plasma total Mo PK parameters was assessed using analysis of variance (ANOVA) statistical model with dosing period, treatment, and treatment sequence as the fixed effects and the participant (sequence) as a random effect, using the natural logarithms of the data; Test type: Other; Geometric Least Square Mean Ratio (%) = 95.0, 90% CI 2-sided [82.1 to 110.0]

2. Primary Outcome: Two-way Crossover Period: Cmax for PUF Mo
Description: Whole blood samples were collected for the measurement of plasma concentrations of PUF Mo via ICP-MS.
Time Frame: predose (0.5 hour) and up to 336 hours postdose
Population: The PKDS-CO included all participants who received at least 1 dose of ALXN1840 in the Two-way Crossover Periods and had evaluable PK data for total and/or PUF molybdenum (as surrogate measures of ALXN1840 PK) in plasma.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Crossover: ALXN1840 Test Formulation (Treatment A) | Crossover: ALXN1840 Reference Formulation (Treatment B)
Number analyzed (Participants) | 46 | 46
ng/mL | 11.758 (43.7) | 12.120 (40.7)
Statistical Analysis 1: Comparison: Crossover: ALXN1840 Test Formulation (Treatment A) vs Crossover: ALXN1840 Reference Formulation (Treatment B); The formulation impact (12 × 1.25 mg EC mini-tablet versus 1 × 15 mg EC tablet) on plasma total Mo PK parameters was assessed using ANOVA statistical model with dosing period, treatment, and treatment sequence as the fixed effects and the participant (sequence) as a random effect, using the natural logarithms of the data; Test type: Other; Geometric Least Square Mean Ratio (%) = 96.243, 90% CI 2-sided [86.384 to 107.227]

3. Primary Outcome: Two-way Crossover Period: Area Under The Plasma Concentration Versus Time Curve From Time 0 To The Last Quantifiable Concentration (AUCt) For Plasma Total Mo
Description: Whole blood samples were collected for the measurement of plasma concentrations of total Mo via ICP-MS.
Time Frame: predose (0.5 hour) and up to 336 hours postdose
Population: The PKDS-CO included all participants who received at least 1 dose of ALXN1840 in the Two-way Crossover Periods and had evaluable PK data for total and/or PUF molybdenum (as surrogate measures of ALXN1840 PK) in plasma. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | Crossover: ALXN1840 Test Formulation (Treatment A) | Crossover: ALXN1840 Reference Formulation (Treatment B)
Number analyzed (Participants) | 45 | 46
hours*ng/mL | 8654.3114 (46.6) | 9253.7266 (44.6)
Statistical Analysis 1: Comparison: Crossover: ALXN1840 Test Formulation (Treatment A) vs Crossover: ALXN1840 Reference Formulation (Treatment B); [analysis description as in outcome 2, analysis 1]; Test type: Other; Geometric Least Square Mean Ratio (%) = 94.9, 90% CI 2-sided [81.6 to 110.5]

4. Primary Outcome: Two-way Crossover Period: AUCt for Plasma PUF Mo
Description: Whole blood samples were collected for the measurement of plasma concentrations of PUF Mo via ICP-MS.
Time Frame: predose (0.5 hour) and up to 336 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | Crossover: ALXN1840 Test Formulation (Treatment A) | Crossover: ALXN1840 Reference Formulation (Treatment B)
Number analyzed (Participants) | 46 | 46
hours*ng/mL | 766.7655 (25.6) | 811.7275 (27.2)
Statistical Analysis 1: Comparison: Crossover: ALXN1840 Test Formulation (Treatment A) vs Crossover: ALXN1840 Reference Formulation (Treatment B); [analysis description as in outcome 2, analysis 1]; Test type: Other; Geometric Least Square Mean Ratio (%) = 101.2, 90% CI 2-sided [70.6 to 145.1]

5. Primary Outcome: Two-way Crossover Period: Area Under The Plasma Concentration Versus Time Curve From Time 0 To Infinity (AUCinf) For Plasma Total Mo
Description: Whole blood samples were collected for the measurement of plasma concentrations of total Mo via ICP-MS.
Time Frame: predose (0.5 hour) and up to 336 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | Crossover: ALXN1840 Test Formulation (Treatment A) | Crossover: ALXN1840 Reference Formulation (Treatment B)
Number analyzed (Participants) | 32 | 35
hours*ng/mL | 10149.7531 (29.2) | 10068.8862 (23.0)
Statistical Analysis 1: Comparison: Crossover: ALXN1840 Test Formulation (Treatment A) vs Crossover: ALXN1840 Reference Formulation (Treatment B); [analysis description as in outcome 2, analysis 1]; Test type: Other; Geometric Least Square Mean Ratio (%) = 99.1, 90% CI 2-sided [89.3 to 109.9]

6. Secondary Outcome: Dose-Proportionality Extension Period: Cmax For Plasma Total Mo
Description: Whole blood samples were collected for the measurement of plasma concentrations of total Mo via ICP-MS.
Time Frame: predose (0.5 hour) and up to 336 hours postdose
Population: The Pharmacokinetic/Pharmacodynamic Set for the Dose-Proportionality Extension Period (PKDS-E) included all participants who receive at least 1 dose of ALXN1840 in the Dose-Proportionality Extension Period and had evaluable PK data for total and/or PUF molybdenum (as surrogate measures of ALXN1840 PK) in plasma.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose-proportionality Extension: ALXN1840 2.5 mg (Treatment C) | Dose-proportionality Extension: ALXN1840 5 mg (Treatment D) | Dose-proportionality Extension: ALXN1840 10 mg (Treatment E) | Dose-proportionality Extension: ALXN1840 30 mg (Treatment F)
Number analyzed (Participants) | 10 | 11 | 9 | 11
ng/mL | 41.0441 (19.48739) | 104.4313 (52.55264) | 199.4759 (55.17849) | 396.0000 (190.18412)

7. Secondary Outcome: Dose-Proportionality Extension Period: Cmax For Plasma PUF Mo
Description: Whole blood samples were collected for the measurement of plasma concentrations of PUF Mo via ICP-MS.
Time Frame: predose (0.5 hour) and up to 336 hours postdose
Population: The PKDS-E included all participants who receive at least 1 dose of ALXN1840 in the Dose-Proportionality Extension Period and had evaluable PK data for total and/or PUF molybdenum (as surrogate measures of ALXN1840 PK) in plasma.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose-proportionality Extension: ALXN1840 2.5 mg (Treatment C) | Dose-proportionality Extension: ALXN1840 5 mg (Treatment D) | Dose-proportionality Extension: ALXN1840 10 mg (Treatment E) | Dose-proportionality Extension: ALXN1840 30 mg (Treatment F)
Number analyzed (Participants) | 10 | 11 | 9 | 11
ng/mL | 8.505 (9.3638) | 9.341 (11.6589) | 16.557 (20.7835) | 25.945 (11.0632)

8. Secondary Outcome: Dose-Proportionality Extension Period: AUCt For Plasma Total Mo
Description: Whole blood samples were collected for the measurement of plasma concentrations of total Mo via ICP-MS.
Time Frame: predose (0.5 hour) and up to 336 hours postdose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | Dose-proportionality Extension: ALXN1840 2.5 mg (Treatment C) | Dose-proportionality Extension: ALXN1840 5 mg (Treatment D) | Dose-proportionality Extension: ALXN1840 10 mg (Treatment E) | Dose-proportionality Extension: ALXN1840 30 mg (Treatment F)
Number analyzed (Participants) | 10 | 11 | 9 | 11
hours*ng/mL | 1677.8616 (736.42903) | 4053.6004 (1601.44215) | 7439.1004 (2213.01844) | 16778.1770 (4707.76069)

9. Secondary Outcome: Dose-Proportionality Extension Period: AUCt For Plasma PUF Mo
Description: Whole blood samples were collected for the measurement of plasma concentrations of PUF Mo via ICP-MS.
Time Frame: predose (0.5 hour) and up to 336 hours postdose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | Dose-proportionality Extension: ALXN1840 2.5 mg (Treatment C) | Dose-proportionality Extension: ALXN1840 5 mg (Treatment D) | Dose-proportionality Extension: ALXN1840 10 mg (Treatment E) | Dose-proportionality Extension: ALXN1840 30 mg (Treatment F)
Number analyzed (Participants) | 10 | 11 | 9 | 11
hours*ng/mL | 584.5782 (177.03965) | 826.2629 (623.23702) | 805.6937 (449.64768) | 976.4214 (220.56479)

10. Secondary Outcome: Dose-Proportionality Extension Period: AUCinf For Plasma Total Mo
Description: Whole blood samples were collected for the measurement of plasma concentrations of total Mo via ICP-MS.
Time Frame: predose (0.5 hour) and up to 336 hours postdose
Population: The PKDS-E included all participants who receive at least 1 dose of ALXN1840 in the Dose-Proportionality Extension Period and had evaluable PK data for total and/or PUF molybdenum (as surrogate measures of ALXN1840 PK) in plasma. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. Only data for Treatments D, E, and F were collected for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | Dose-proportionality Extension: ALXN1840 5 mg (Treatment D) | Dose-proportionality Extension: ALXN1840 10 mg (Treatment E) | Dose-proportionality Extension: ALXN1840 30 mg (Treatment F)
Number analyzed (Participants) | 6 | 6 | 10
hours*ng/mL | 4920.5103 (1035.21136) | 9057.1367 (1345.89511) | 17842.1736 (5496.94190)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 15
Description: The Safety Set included all participants who received at least 1 dose of ALXN1840 and are presented by the treatment received at the time of the adverse event reporting.
Groups:
- Dose-proportionality Extension: ALXN1840 5 mg (Treatment D: Participants received a single dose of ALXN1840 5 mg (4 × 1.25 mg EC mini-tablets) orally on Day 1.
Arm/Group | Crossover: ALXN1840 Test Formulation (Treatment A) | Crossover: ALXN1840 Reference Formulation (Treatment B) | Dose-proportionality Extension: ALXN1840 2.5 mg (Treatment C) | Dose-proportionality Extension: ALXN1840 5 mg (Treatment D | Dose-proportionality Extension: ALXN1840 10 mg (Treatment E) | Dose-proportionality Extension: ALXN1840 30 mg (Treatment F)
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/46 | 0/10 | 0/11 | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46 | 0/10 | 0/11 | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 18/46 | 20/46 | 2/10 | 5/11 | 3/9 | 4/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crossover: ALXN1840 Test Formulation (Treatment A) (N=46) | Crossover: ALXN1840 Reference Formulation (Treatment B) (N=46) | Dose-proportionality Extension: ALXN1840 2.5 mg (Treatment C) (N=10) | Dose-proportionality Extension: ALXN1840 5 mg (Treatment D (N=11) | Dose-proportionality Extension: ALXN1840 10 mg (Treatment E) (N=9) | Dose-proportionality Extension: ALXN1840 30 mg (Treatment F) (N=11)
Headache (Nervous system disorders) | 6 | 3 | 1 | 1 | 2 | 2
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 1 | 3 | 0 | 0 | 0 | 0
Catheter site bruise (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Catheter site paraesthesia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Feeling abnormal (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Feeling abnormal (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vessel puncture site reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 0 | 0 | 0 | 0 | 0
Premenstrual pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site thrombosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Physical deconditioning (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tonsillolith (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Monocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/80/NCT04610580/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT04610580/SAP_001.pdf